CLINICAL TRIAL: NCT01105611
Title: An Open-label, Randomised Pilot Study Comparing the Efficacy, Safety and Tolerability of Raltegravir With Protease Inhibitor-based Therapy in Treatment-naïve, HIV/Hepatitis C Co-infected Injecting Drug Users Receiving Methadone
Brief Title: Safety and Efficacy Study Comparing Raltegravir to a Protease Inhibitor in Treatment-naïve, HIV/Hepatitis C Drug Users
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: St. James's Hospital, Ireland (Other)
Responsible Party: Professor Colm Bergin, St. James's Hospital, Dublin, Ireland
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CB-2010-01; 2010-018326-39 (EudraCT Number)
Record Dates: First submitted 2010-04-14; First posted 2010-04-16 (Estimated); Last update posted 2011-07-21 (Estimated); Status verified 2010-03

CONDITIONS: HIV Infections; Hepatitis C
Keywords: HIV; Hepatitis C; Co-infection; Intravenous drug users; Treatment-naïve; Methadone
MeSH Terms: conditions — HIV Infections; Hepatitis C; Coinfection | interventions — Raltegravir Potassium; atazanavir, ritonavir drug combination; Atazanavir Sulfate; Ritonavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Raltegravir (Experimental): Raltegravir in combination with Tenofovir/Emtricitabine
  Interventions: Drug: Raltegravir
- Atazanavir/Ritonavir (Active Comparator): Atazanavir 300mg orally once daily with Ritonavir 100mg orally once daily; together with combination of Tenofovir/Emtricitabine
  Interventions: Drug: Atazanavir/Ritonavir

INTERVENTIONS:
Drug: Raltegravir — 400mg orally twice daily. Number of cycles: unless toxicity or treatment failure occurs, there will be no anticipated treatment discontinuation.
  Other Names: Isentress™
  Arms: Raltegravir
Drug: Atazanavir/Ritonavir — Atazanavir 300mg orally once daily boosted with Ritonavir orally 100mg once daily. Number of cycles: unless toxicity or treatment failure occurs, there will be no anticipated treatment discontinuation.
  Other Names: Reyataz™ (Atazanavir), Norvir™ (Ritonavir)
  Arms: Atazanavir/Ritonavir

SUMMARY:
The purpose of this study is to compare how safe, tolerable, and effective a novel drug, raltegravir, is to a commonly used combination, atazanavir/ritonavir, as initial treatment in HIV/Hepatitis C co-infected injecting drug users on a methadone program.

DETAILED DESCRIPTION:
Raltegravir is an HIV-1 integrase inhibitor that is currently licensed for use in treatment-experienced HIV-1 patients and recently approved for use in treatment-naïve patients. Recent data has shown that the virologic response in patients on raltegravir with no history of antiretroviral treatment (ART) was equal to efavirenz-based therapy at 96-weeks (combined with tenofovir/lamivudine). Moreover, raltegravir demonstrated greater immunologic effect, had fewer adverse side effects and had a neutral effect on lipid levels. Further support for first-line use comes from recent 48-week data of a subgroup analyses of the STARTMRK Phase III study comparing raltegravir to efavirenz-based therapy (with tenofovir/emtricitabine) in treatment-naïve patients that showed non-inferior virologic and immunologic efficacy with raltegravir. There were significantly fewer overall and drug-related clinical adverse events in the raltegravir group and a similar safety profile in patients with hepatitis B and/or C co-infection. These findings suggest that use of raltegravir as a component of initial therapy might be beneficial in patients with significant co-morbidities such as hepatitis C and in situations where there is concern of interactions between antiretrovirals and other drugs.

Injecting drug users (IDUs) represent a patient group where there are formidable challenges in HIV treatment. Difficulties in management arise not only from substance abuse but also because of high rates of social instability and psychiatric co-morbidities. Furthermore, many in this patient group have hepatitis C co-infection. These confounding factors negatively impact adherence to, and ultimately the efficacy of treatment and can affect physician perception when prescribing antiretrovirals. Concurrent methadone therapy further complicates HIV treatment because of its potential side effects and interactions with antiretrovirals. However, methadone maintenance therapy also represents an important opportunity to engage patients in consistent medical care and has been shown to improve adherence to antiretroviral treatment and thus viral suppression.

The incidence of co-infection with HIV and hepatitis C virus (HCV) in IDUs is high. An estimated 50-90% of IDUs in the U.S. are co-infected with HIV/Hepatitis C according to the Center for Disease Control and Prevention. HIV co-infection aggravates the natural course of HCV infection. In a meta-analysis of the effect of HIV on the progression of HCV liver disease compared to mono-infection with HCV, the relative risk of end-stage liver disease (ESLD) and cirrhosis with HIV co-infection was found to be 6.14 and 2.07, respectively. Difficulties arise in the treatment of HIV with respect to HCV liver disease. Drug hepatotoxicity is a major concern in the selection of an appropriate antiretroviral regimen. Optimising therapy in this patient group necessitates a balance between retroviral suppression and minimising hepatic side effects.

Raltegravir is predominantly metabolised by hepatic glucuronidation via the uridine diphosphate glucuronosyltransferase 1A1 (UGT1A1) isozyme. A small component is renally excreted (~9%). In three double-blind, randomised studies of pharmacokinetics, safety and tolerability, raltegravir was found to be rapidly absorbed with a terminal half-life of 7-12 hours. It exhibited potent in vitro inhibition with a 95% inhibitory concentration (IC95) = 33nM in 50% human serum. Pharmacokinetic analyses of various dosing regimens supported the use of twice daily dosing of multiple doses of 100mg and greater. Results from a study investigating once daily dosing are pending.

Hepatic impairment is less likely to affect UGT1A1 metabolism in comparison to other liver metabolic pathways. A recent study evaluated the effect of liver impairment on raltegravir pharmacokinetics in 20 HIV-negative patients (ten patients with moderate hepatic insufficiency and ten healthy, matched controls). The geometric mean ratios (GMR: mean value for the group with moderate hepatic insufficiency/mean value for the healthy controls) and 90% confidence intervals (CIs) for the area under the concentration-time curve from time zero to infinity (AUC0- ∞ ), the maximum concentration of drug in plasma (Cmax), and the concentration at 12 h (C12) were 0.86 (90% CI, 0.41, 1.77), 0.63 (90% CI, 0.23, 1.70), and 1.26 (90% CI, 0.65, 2.43), respectively. The study authors determined that liver impairment produced no clinically significant effects on raltegravir pharmacokinetics and therefore no dose adjustments are needed for mild to moderate hepatic insufficiency.

Protease inhibitors, such as atazanavir, are extensively metabolised via hepatic cytochrome P450 (CYP) 3A isozymes. In patients with hepatic insufficiency, dose adjustments of PIs or consideration of alternative therapies may be necessary. Atazanavir is also a potent inhibitor of CYP3A and therefore has a potential to cause drug interactions .

Concerns regarding adverse cardiac effects of antiretroviral therapy have recently emerged. Protease inhibitors have been associated with an increased risk of myocardial infarction that is partially due to dyslipidaemia. Ritonavir-boosted atazanavir is commonly used as part of combination treatment in IDUs because of its modest effect on lipid levels and also due to the simplicity of once daily dosing. However, it has other associated risk factors and intolerability due to hyperbilirubinaemia is also an issue.

There is also growing concern with reports of long QT syndrome and torsade de pointes in IDUs. This patient group have several risk factors that increase their susceptibility. Methadone is well recognised to cause long QT syndrome and torsades de pointes through inhibition of a cardiac potassium channel, the major component of which is encoded by the human ether-a-go-go gene (HERG). Multiple HERG polymorphisms have been identified that are clinically silent but may confer vulnerability to arrhythmia by a triggering event. Protease inhibitors also have the potential to cause QT prolongation. This may be mediated by direct effects on HERG channels or by potentiating the effects of other drugs through inhibition of CYP3A, or both. Concurrent use of protease inhibitors and methadone might pose an additive risk of QT prolongation and a few cases have been reported recently. Additionally, co-infection with hepatitis C is also recognised to prolong the QT interval.

Raltegravir has been shown to have no effect on the QT interval in a single, supratherapeutic dose in humans and in multiple doses in an animal model. It also exhibits negligible inhibition of HERG current in vitro and has been found to have little to no effect on cytochrome P450 enzymes.

In summary, efficacious virologic and immunologic response, safe use in hepatic impairment, non-inhibition of CYP enzymes, lack of QT effect, and favourable lipid and side effect profile indicate that raltegravir could be a preferred option for first-line treatment in this patient group.

This study will be carried out as a Phase 4, Multi-Centre Open Label, Investigator Led, Randomised Pilot Study to compare the efficacy, safety and tolerability of raltegravir (Isentress™) with protease inhibitor-based therapy atazanavir/ritonavir (Reyataz™/Norvir™) in treatment naïve, HIV/Hepatitis C co-infected injecting drug users receiving methadone. Patients who are attending a drug treatment clinic, who are on methadone maintenance therapy, who fulfill standard criteria to receive antiretroviral therapy (ART) and who meet all other study specific eligibility criteria will be invited to participate in the study.

Eligible patients, who are willing to participate in the study and who agree to comply with all study treatments and procedures, will be randomized to treatment with either:

1. Raltegravir 400mg PO twice daily; or
2. Atazanavir/ritonavir 300mg/100mg PO once daily over a 96 week treatment period.

As per the recommended guidelines, both treatment regimes will be combined with a nucleoside reverse-transcriptase inhibitor (NRTI) backbone of tenofovir and emtricitabine, but can be changed due to toxicities as per the discretion of the investigator or other medically qualified designee.

The total study duration for subjects completing the entire study will be approximately 100 weeks. During this time subjects will attend the clinic for 11 study visits at Baseline, Weeks 4, 12, 24, 36, 48, 60, 72, 84 and 96 and an End of Study Visit, 4 weeks post completion of treatment.

Subjects' participation in this study will end following the End of Study Visit (or early withdrawal visit if applicable). Once subjects have completed their participation in this study they will be treated as per routine standard care for this patient population.

Written informed consent will be obtained prior to any study procedures being conducted. Patients will have an initial baseline assessment prior to treatment initiation. This will include a medical history, physical examination and electrocardiogram. Baseline laboratory tests will include a resistance profile, CD4 count, viral load, hepatitis C status, full blood count, liver blood tests and renal profile.

Patients will be re-assessed at 4, 12, 24, 36, 48, 60, 72, 84 and 96 weeks post initiation for treatment efficacy, safety, tolerability and compliance. Follow-up blood tests will be drawn to assess virological and immunological response to treatment as well as routine blood tests to detect hepatitis C status, liver/renal toxicities and haematological abnormalities. ECG evaluation for QT abnormalities will be performed at baseline and at weeks 4, 12, 48 and 96. A follow up safety visit will be conducted 4 weeks post completion of therapy. Monitoring for adverse events will take place throughout the study period and continuity of care, as per standard medical care for this patient population, maintained after the patients have completed the study at the respective sites.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female Patients Age ≥ 18 years old.
* Naïve to antiretroviral treatment.
* Subject must be willing and able to understand and provide written, informed consent prior to participation in the study.
* Subjects must be on concurrent methadone maintenance therapy.
* Documented HIV infection (antibody positive).
* Documented Hepatitis C co-infection (PCR positive).
* HIV RNA > 5,000.
* Indication for starting ART according to guidelines.
* Documented resistance profile taken at baseline and includes investigational medicinal products.
* Females may be eligible for enrolment in the study if she is of:

  1. Non-childbearing potential; or, Child-bearing potential females must have a negative pregnancy test at initial screening and agree to an acceptable barrier and/or hormonal method of contraception; Sterilization

Exclusion Criteria:

* Subject is in the initial acute phase of a CDC Clinical Category C infection at Baseline. Subjects may be enrolled provided they are receiving treatment for such infections and are clinically improving at the Baseline visit.
* Concurrent treatment with an investigational drug or participation in another clinical trial.
* Use of an investigational drug within 4 weeks or 5 half-lives, whichever is longer, preceding the first dose of investigational medicinal product.
* Subject is, in the opinion of the investigator, unable to complete the study dosing period and protocol evaluations and assessments.
* Subject has evidence of genotypic (as defined by the current ANRS AC-11 algorithm) resistance to raltegravir, atazanavir and ritonavir at screening.
* Patients with alcohol and drug use problems that in the view of investigator will compromise participation in the study.
* Elevated alanine aminotransferase (ALT) > 5 times upper limit of normal (ULN)
* Subjects with severe hepatic impairment (Child-Pugh score > 9).
* Subjects receiving treatment for HCV.
* Subjects with concurrent HBV infection.
* Subject is pregnant or breast feeding.
* Subject suffers from any serious medical condition which would compromise the safety of the subject.
* Subject has a pre-existing mental, physical, or substance abuse disorder that may interfere with the subject's ability to comply with the dosing schedule and protocol evaluations and assessments.
* Subject has a condition or disorder which may interfere with drug absorption or render the subject unable to take oral medication.
* Subject has any acute laboratory abnormality at screening, which, in the opinion of the Investigator, would preclude the subject's participation in the study of an investigational compound. Any verified Grade 4 laboratory abnormality would exclude a subject from study participation.
* Subject has an estimated creatinine clearance < 50 mL/min via the Cockcroft-Gault method [Cockcroft, 1976].
* Subject is receiving, or has received within 14 days prior to screen, any drug that has been classified as 'contraindicated' from use with RAL or ATV/RTV.
* Subject has received treatment with radiation therapy or cytotoxic chemotherapeutic agents within 28 days prior to Screening, or has an anticipated need for these agents within the study period.
* Subject has received treatment with an HIV-1 immunotherapeutic vaccine or any agents with documented activity against HIV-1 in vitro within 28 days prior to screening, or an anticipated need during the study.
* Subjects who require treatment with any contraindicated medications within 14 days of commencement of investigational medicinal product, or an anticipated need during the study.
* Subject has a history of allergy to any of the investigational medicinal products or any excipients therein.
* Subject has prolonged QTc interval on screening electrocardiogram (repeated demonstration of a QTc interval >450ms in men and >470ms in women).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2010-08; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of grade 3-4 liver function test (LFT) elevations | 4 weeks
Incidence of grade 3-4 liver function test (LFT) elevations | 12 weeks
Incidence of grade 3-4 liver function test (LFT) elevations | 24 weeks
Incidence of grade 3-4 liver function test (LFT) elevations | 36 weeks
Incidence of grade 3-4 liver function test (LFT) elevations | 48 weeks
Incidence of grade 3-4 liver function test (LFT) elevations | 60 weeks
Incidence of grade 3-4 liver function test (LFT) elevations | 72 weeks
Incidence of grade 3-4 liver function test (LFT) elevations | 84 weeks
Incidence of grade 3-4 liver function test (LFT) elevations | 96 weeks
Viral suppression | 24 weeks
  Viral suppression is defined as HIV-1 RNA less than 50 copies per mL

SECONDARY OUTCOMES:
Viral suppression | 48 weeks
  Viral suppression is defined as HIV- RNA less than 50 copies per mL.
Immunologic response | 96 weeks
  Recovery of CD4 count
Overall safety in patients with mild to moderate hepatic impairment | 48 weeks
Outpatient retention rates | 96 weeks
QTc interval changes | 4 weeks
  Effects of pharmacological intervention on corrected QT interval on electrocardiogram
Immunologic response | 24 weeks
Immunologic response | 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Colm Bergin, MD, FRCPI, Principal Investigator — Department of Genitourinary Medicine and Infectious Diseases, St. James's Hospital, Dublin, Ireland
Locations (2):
- Ireland (2):
  - Department of Genitourinary Medicine and Infectious Diseases, St. James's Hospital, Dublin
  - Mater Misericordiae University Hospital, Dublin

REFERENCES:
- [Background] Markowitz M, Nguyen BY, Gotuzzo E, Mendo F, Ratanasuwan W, Kovacs C, Prada G, Morales-Ramirez JO, Crumpacker CS, Isaacs RD, Campbell H, Strohmaier KM, Wan H, Danovich RM, Teppler H; Protocol 004 Part II Study Team. Sustained antiretroviral effect of raltegravir after 96 weeks of combination therapy in treatment-naive patients with HIV-1 infection. J Acquir Immune Defic Syndr. 2009 Nov 1;52(3):350-6. doi: 10.1097/QAI.0b013e3181b064b0. PMID 19648823
- [Background] Lennox JL, DeJesus E, Lazzarin A, Pollard RB, Madruga JV, Berger DS, Zhao J, Xu X, Williams-Diaz A, Rodgers AJ, Barnard RJ, Miller MD, DiNubile MJ, Nguyen BY, Leavitt R, Sklar P; STARTMRK investigators. Safety and efficacy of raltegravir-based versus efavirenz-based combination therapy in treatment-naive patients with HIV-1 infection: a multicentre, double-blind randomised controlled trial. Lancet. 2009 Sep 5;374(9692):796-806. doi: 10.1016/S0140-6736(09)60918-1. Epub 2009 Aug 3. PMID 19647866
- [Background] O'Connor PG, Selwyn PA, Schottenfeld RS. Medical care for injection-drug users with human immunodeficiency virus infection. N Engl J Med. 1994 Aug 18;331(7):450-9. doi: 10.1056/NEJM199408183310707. No abstract available. PMID 8035842
- [Background] Waldrop-Valverde D, Valverde E. Homelessness and psychological distress as contributors to antiretroviral nonadherence in HIV-positive injecting drug users. AIDS Patient Care STDS. 2005 May;19(5):326-34. doi: 10.1089/apc.2005.19.326. PMID 15916495
- [Background] Lucas GM, Cheever LW, Chaisson RE, Moore RD. Detrimental effects of continued illicit drug use on the treatment of HIV-1 infection. J Acquir Immune Defic Syndr. 2001 Jul 1;27(3):251-9. doi: 10.1097/00126334-200107010-00006. PMID 11464144
- [Background] Lucas GM, Griswold M, Gebo KA, Keruly J, Chaisson RE, Moore RD. Illicit drug use and HIV-1 disease progression: a longitudinal study in the era of highly active antiretroviral therapy. Am J Epidemiol. 2006 Mar 1;163(5):412-20. doi: 10.1093/aje/kwj059. Epub 2006 Jan 4. PMID 16394200
- [Background] Lucas GM, Mullen BA, Weidle PJ, Hader S, McCaul ME, Moore RD. Directly administered antiretroviral therapy in methadone clinics is associated with improved HIV treatment outcomes, compared with outcomes among concurrent comparison groups. Clin Infect Dis. 2006 Jun 1;42(11):1628-35. doi: 10.1086/503905. Epub 2006 Apr 28. PMID 16652321
- [Background] Graham CS, Baden LR, Yu E, Mrus JM, Carnie J, Heeren T, Koziel MJ. Influence of human immunodeficiency virus infection on the course of hepatitis C virus infection: a meta-analysis. Clin Infect Dis. 2001 Aug 15;33(4):562-9. doi: 10.1086/321909. Epub 2001 Jul 6. PMID 11462196
- [Background] Kassahun K, McIntosh I, Cui D, Hreniuk D, Merschman S, Lasseter K, Azrolan N, Iwamoto M, Wagner JA, Wenning LA. Metabolism and disposition in humans of raltegravir (MK-0518), an anti-AIDS drug targeting the human immunodeficiency virus 1 integrase enzyme. Drug Metab Dispos. 2007 Sep;35(9):1657-63. doi: 10.1124/dmd.107.016196. Epub 2007 Jun 25. PMID 17591678
- [Background] Iwamoto M, Wenning LA, Petry AS, Laethem M, De Smet M, Kost JT, Merschman SA, Strohmaier KM, Ramael S, Lasseter KC, Stone JA, Gottesdiener KM, Wagner JA. Safety, tolerability, and pharmacokinetics of raltegravir after single and multiple doses in healthy subjects. Clin Pharmacol Ther. 2008 Feb;83(2):293-9. doi: 10.1038/sj.clpt.6100281. Epub 2007 Aug 22. PMID 17713476
- [Background] Furlan V, Demirdjian S, Bourdon O, Magdalou J, Taburet AM. Glucuronidation of drugs by hepatic microsomes derived from healthy and cirrhotic human livers. J Pharmacol Exp Ther. 1999 May;289(2):1169-75. PMID 10215701
- [Background] Iwamoto M, Hanley WD, Petry AS, Friedman EJ, Kost JT, Breidinger SA, Lasseter KC, Robson R, Lunde NM, Wenning LA, Stone JA, Wagner JA. Lack of a clinically important effect of moderate hepatic insufficiency and severe renal insufficiency on raltegravir pharmacokinetics. Antimicrob Agents Chemother. 2009 May;53(5):1747-52. doi: 10.1128/AAC.01194-08. Epub 2009 Feb 17. PMID 19223645
- [Background] Le Tiec C, Barrail A, Goujard C, Taburet AM. Clinical pharmacokinetics and summary of efficacy and tolerability of atazanavir. Clin Pharmacokinet. 2005;44(10):1035-50. doi: 10.2165/00003088-200544100-00003. PMID 16176117
- [Background] Perloff ES, Duan SX, Skolnik PR, Greenblatt DJ, von Moltke LL. Atazanavir: effects on P-glycoprotein transport and CYP3A metabolism in vitro. Drug Metab Dispos. 2005 Jun;33(6):764-70. doi: 10.1124/dmd.104.002931. Epub 2005 Mar 11. PMID 15764714
- [Background] Friis-Moller N, Sabin CA, Weber R, d'Arminio Monforte A, El-Sadr WM, Reiss P, Thiebaut R, Morfeldt L, De Wit S, Pradier C, Calvo G, Law MG, Kirk O, Phillips AN, Lundgren JD; Data Collection on Adverse Events of Anti-HIV Drugs (DAD) Study Group. Combination antiretroviral therapy and the risk of myocardial infarction. N Engl J Med. 2003 Nov 20;349(21):1993-2003. doi: 10.1056/NEJMoa030218. PMID 14627784
- [Background] DAD Study Group; Friis-Moller N, Reiss P, Sabin CA, Weber R, Monforte Ad, El-Sadr W, Thiebaut R, De Wit S, Kirk O, Fontas E, Law MG, Phillips A, Lundgren JD. Class of antiretroviral drugs and the risk of myocardial infarction. N Engl J Med. 2007 Apr 26;356(17):1723-35. doi: 10.1056/NEJMoa062744. PMID 17460226
- [Background] Ehret GB, Voide C, Gex-Fabry M, Chabert J, Shah D, Broers B, Piguet V, Musset T, Gaspoz JM, Perrier A, Dayer P, Desmeules JA. Drug-induced long QT syndrome in injection drug users receiving methadone: high frequency in hospitalized patients and risk factors. Arch Intern Med. 2006 Jun 26;166(12):1280-7. doi: 10.1001/archinte.166.12.1280. PMID 16801510
- [Background] Krantz MJ, Lewkowiez L, Hays H, Woodroffe MA, Robertson AD, Mehler PS. Torsade de pointes associated with very-high-dose methadone. Ann Intern Med. 2002 Sep 17;137(6):501-4. doi: 10.7326/0003-4819-137-6-200209170-00010. PMID 12230351
- [Background] Katchman AN, McGroary KA, Kilborn MJ, Kornick CA, Manfredi PL, Woosley RL, Ebert SN. Influence of opioid agonists on cardiac human ether-a-go-go-related gene K(+) currents. J Pharmacol Exp Ther. 2002 Nov;303(2):688-94. doi: 10.1124/jpet.102.038240. PMID 12388652
- [Background] Anson BD, Ackerman MJ, Tester DJ, Will ML, Delisle BP, Anderson CL, January CT. Molecular and functional characterization of common polymorphisms in HERG (KCNH2) potassium channels. Am J Physiol Heart Circ Physiol. 2004 Jun;286(6):H2434-41. doi: 10.1152/ajpheart.00891.2003. Epub 2004 Feb 19. PMID 14975928
- [Background] Anson BD, Weaver JG, Ackerman MJ, Akinsete O, Henry K, January CT, Badley AD. Blockade of HERG channels by HIV protease inhibitors. Lancet. 2005 Feb 19-25;365(9460):682-6. doi: 10.1016/S0140-6736(05)17950-1. PMID 15721475
- [Background] Ly T, Ruiz ME. Prolonged QT interval and torsades de pointes associated with atazanavir therapy. Clin Infect Dis. 2007 Mar 15;44(6):e67-8. doi: 10.1086/511875. Epub 2007 Feb 1. PMID 17304444
- [Background] Josephson F, Bertilsson L, Bottiger Y, Flamholc L, Gisslen M, Ormaasen V, Sonnerborg A, Diczfalusy U. CYP3A induction and inhibition by different antiretroviral regimens reflected by changes in plasma 4beta-hydroxycholesterol levels. Eur J Clin Pharmacol. 2008 Aug;64(8):775-81. doi: 10.1007/s00228-008-0492-8. Epub 2008 May 6. PMID 18458892
- [Background] Gallagher DP, Kieran J, Sheehan G, Lambert J, Mahon N, Mallon PW. Ritonavir-boosted atazanavir, methadone, and ventricular tachycardia: 2 case reports. Clin Infect Dis. 2008 Aug 1;47(3):e36-8. doi: 10.1086/589869. PMID 18558878
- [Background] Nordin C, Kohli A, Beca S, Zaharia V, Grant T, Leider J, Marantz P. Importance of hepatitis C coinfection in the development of QT prolongation in HIV-infected patients. J Electrocardiol. 2006 Apr;39(2):199-205. doi: 10.1016/j.jelectrocard.2005.09.001. Epub 2005 Nov 28. PMID 16580420
- [Background] Iwamoto M, Kost JT, Mistry GC, Wenning LA, Breidinger SA, Marbury TC, Stone JA, Gottesdiener KM, Bloomfield DM, Wagner JA. Raltegravir thorough QT/QTc study: a single supratherapeutic dose of raltegravir does not prolong the QTcF interval. J Clin Pharmacol. 2008 Jun;48(6):726-33. doi: 10.1177/0091270008318007. Epub 2008 Apr 25. PMID 18441333